CLINICAL TRIAL: NCT05333640
Title: A Real-world Registry Investigating Sirolimus-coated Balloon Versus Paclitaxel-coated Balloon Angioplasty for the Treatment of Dysfunctional Arteriovenous Fistula
Acronym: SAVE AVF
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Singapore General Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 2022/2014
Record Dates: First submitted 2022-04-11; First posted 2022-04-19 (Actual); Last update posted 2022-04-19 (Actual); Status verified 2022-04

CONDITIONS: Dialysis Access Malfunction; Stenosis
MeSH Terms: conditions — Constriction, Pathologic

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- AVFs treated with Sirolimus Drug Coated Balloon: Dysfunctional matured AVF that have underwent thrombolysis or balloon angioplasty with SDCB within 6 months witll be considered for the registry.
  Interventions: Device: Sirolimus Drug Coated Balloon
- AVFs treated with Paclitaxel Drug Coated Balloon: Dysfunctional matured AVF that have underwent thrombolysis or balloon angioplasty with PDCB within 6 months witll be considered for the registry.
  Interventions: Device: Paclitaxel Drug Coated Balloon

INTERVENTIONS:
Device: Sirolimus Drug Coated Balloon — AVFs treated with SDCB
  Groups: AVFs treated with Sirolimus Drug Coated Balloon
Device: Paclitaxel Drug Coated Balloon — AVFs treated with PDCB
  Groups: AVFs treated with Paclitaxel Drug Coated Balloon

SUMMARY:
Drug-coated balloon (DCB) angioplasty has been shown to be superior to POBA in the treatment of stenosis in AVF. This is because the very intervention used to treat underlying stenosis by POBA can induce vascular injury and accelerate intimal hyperplasia, resulting in rapid restenosis and need for repeated procedure to maintain vessel patency. The anti-proliferative drug that is coated on the surface of balloon is released to the vessel wall during balloon angioplasty and blunt the acceleration of intimal hyperplasia response, resulting in improved primary patency after angioplasty. Additionally, unlike stents, DCB does not leave a permanent structure that may impede future surgical revision. Recent randomized control trials (RCT) have shown the superiority of paclitaxel durg-coated balloon (PDCB) over POBA in the treatment of stenosis in AVFs. In a large multicenter RCT, PDCB was demonstrated to result in a 6-month target lesion primary patency of 82.2% compared to 59.5% for POBA. However, concerns had also arisen recently in the use of PDCB. In large lower limb studies involving the use of paclitaxel devices, meta-analysis by Katsanos et al had revealed increased late risk mortality in patient that are treated with PDCB or paclitaxel-coated stent.

Sirolimus drug-coated balloon (SDCB) is the new generation of drug eluting balloons that are available in the market. Compared to paclitaxel, sirolimus is cytostatic in its mode of action with a high margin of safety. It has a high transfer rate to the vessel wall and effectively inhibit neointimal hyperplasia in the porcine coronary model. The effectiveness of SDCB in patients with dialysis access dysfunction has been shown in a small pilot study in AVF stenosis and AVG thrombosis. SAVE AVF registry ams to assess the efficacy and safety of SDCB vs PDCB angioplasty.

ELIGIBILITY:
Inclusion Criteria:

* Age 21-85 years
* Patient who required balloon angioplasty for dysfunctional or thrombosed AVF
* Successful thrombolysis and angioplasty of the underlying stenosis, defined as less than 30% residual stenosis on Digital Subtraction Angiography (DSA) based on visual assessment of the operator and restoration of thrill in the AVF on clinical examination. For concurrent asymptomatic or angiographically not significant central vein stenosis, patients can be included in no treatment is required.
* received either PDCB or SDCB for the treatment of stenosis.

Exclusion Criteria:

* Patient unable to provide informed consent
* Presence of symptomatic or angiographically significant central vein stenosis who require treatment, with more than 30% residual stenosis post angioplasty
* Patients who had underwent stent placement within the AVF circuit
* Sepsis or active infection
* Recent intracranial bleed or gastrointestinal bleed within the past 12 months.
* Allergy to iodinated contrast media, heparin, paclitaxel or sirolimus
* Pregnancy
* Inadequate treatment of underlying stenosis, defined as >= 30% residual stenosis of the underlying lesions.

Ages: 21 Years to 85 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients with dysfunctional AVFs who have undergone balloon angioplasty or thrombolysis with PDCB or SDCB.
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2022-04-18 (Estimated); Primary Completion 2023-10-30 (Estimated); Study Completion 2024-04-30 (Estimated)

PRIMARY OUTCOMES:
Circuit Primary Patency Rate at 6 months | 6 months post-op
  Circuit primary patency is lost if patient has to undergo a repeat intervention that is clinically driven. Clinically driven indication may be based on physical examination such as loss of thrill, pulsatile flow or swollen arm.

SECONDARY OUTCOMES:
Circuit Primary Patency at 12 months | 12 months post-op
  Circuit primary patency is lost if patient has to undergo a repeat intervention that is clinically driven. Clinically driven indication may be based on physical examination such as loss of thrill, pulsatile flow or swollen arm.
Target Lesion Restenosis | 6 and 12 months post-op
  Incidence of stenosis >50% diameter of adjacent reference vessel segment from angiography images
Number of repeat interventions to treated lesion | 6 and 12 months post-op
Number of repeat interventions to maintain access circuit | 6 and 12 months post-op
  This will include interventions to treated lesion
Target lesion revascularization free interval | 12 months post-op
  Interval from intervention to repeat clinically driven target lesion reintervention
Complication rates of the procedure | Time of procedure
  Categorised according to SIR definitions (Aruny et al)
Mortality rates of patients | 6 and 12 months post-op

CONTACTS AND LOCATIONS:
Overall Officials: Tjun Tip Tang, Principal Investigator — Singapore General Hospital; Ru Yu Tan, Principal Investigator — Singapore General Hospital; Apoorva Gogna, Principal Investigator — Singapore General Hospital
Locations (1):
- Singapore General Hospital, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Roy-Chaudhury P, Sukhatme VP, Cheung AK. Hemodialysis vascular access dysfunction: a cellular and molecular viewpoint. J Am Soc Nephrol. 2006 Apr;17(4):1112-27. doi: 10.1681/ASN.2005050615. PMID 16565259
- [Background] Lee T, Roy-Chaudhury P. Advances and new frontiers in the pathophysiology of venous neointimal hyperplasia and dialysis access stenosis. Adv Chronic Kidney Dis. 2009 Sep;16(5):329-38. doi: 10.1053/j.ackd.2009.06.009. PMID 19695501
- [Background] Pantelias K, Grapsa E. Vascular access today. World J Nephrol. 2012 Jun 6;1(3):69-78. doi: 10.5527/wjn.v1.i3.69. PMID 24175244
- [Background] Rajan DK, Bunston S, Misra S, Pinto R, Lok CE. Dysfunctional autogenous hemodialysis fistulas: outcomes after angioplasty--are there clinical predictors of patency? Radiology. 2004 Aug;232(2):508-15. doi: 10.1148/radiol.2322030714. PMID 15286321
- [Background] Manninen HI, Kaukanen ET, Ikaheimo R, Karhapaa P, Lahtinen T, Matsi P, Lampainen E. Brachial arterial access: endovascular treatment of failing Brescia-Cimino hemodialysis fistulas--initial success and long-term results. Radiology. 2001 Mar;218(3):711-8. doi: 10.1148/radiology.218.3.r01mr38711. PMID 11230644
- [Background] Heye S, Maleux G, Vaninbroukx J, Claes K, Kuypers D, Oyen R. Factors influencing technical success and outcome of percutaneous balloon angioplasty in de novo native hemodialysis arteriovenous fistulas. Eur J Radiol. 2012 Sep;81(9):2298-303. doi: 10.1016/j.ejrad.2011.09.004. Epub 2011 Sep 28. PMID 21955605
- [Background] Haskal ZJ, Trerotola S, Dolmatch B, Schuman E, Altman S, Mietling S, Berman S, McLennan G, Trimmer C, Ross J, Vesely T. Stent graft versus balloon angioplasty for failing dialysis-access grafts. N Engl J Med. 2010 Feb 11;362(6):494-503. doi: 10.1056/NEJMoa0902045. PMID 20147715
- [Background] Shemesh D, Goldin I, Zaghal I, Berlowitz D, Raveh D, Olsha O. Angioplasty with stent graft versus bare stent for recurrent cephalic arch stenosis in autogenous arteriovenous access for hemodialysis: a prospective randomized clinical trial. J Vasc Surg. 2008 Dec;48(6):1524-31, 1531.e1-2. doi: 10.1016/j.jvs.2008.07.071. Epub 2008 Oct 1. PMID 18829240
- [Background] Salman L, Asif A. Stent graft for nephrologists: concerns and consensus. Clin J Am Soc Nephrol. 2010 Jul;5(7):1347-52. doi: 10.2215/CJN.02380310. Epub 2010 May 27. PMID 20507955
- [Background] Allon M. Current management of vascular access. Clin J Am Soc Nephrol. 2007 Jul;2(4):786-800. doi: 10.2215/CJN.00860207. Epub 2007 May 30. PMID 17699495
- [Background] Katsanos K, Karnabatidis D, Kitrou P, Spiliopoulos S, Christeas N, Siablis D. Paclitaxel-coated balloon angioplasty vs. plain balloon dilation for the treatment of failing dialysis access: 6-month interim results from a prospective randomized controlled trial. J Endovasc Ther. 2012 Apr;19(2):263-72. doi: 10.1583/11-3690.1. PMID 22545894
- [Background] Kennedy SA, Mafeld S, Baerlocher MO, Jaberi A, Rajan DK. Drug-Coated Balloon Angioplasty in Hemodialysis Circuits: A Systematic Review and Meta-Analysis. J Vasc Interv Radiol. 2019 Apr;30(4):483-494.e1. doi: 10.1016/j.jvir.2019.01.012. Epub 2019 Mar 8. PMID 30857987
- [Background] Katsanos K, Spiliopoulos S, Kitrou P, Krokidis M, Karnabatidis D. Risk of Death Following Application of Paclitaxel-Coated Balloons and Stents in the Femoropopliteal Artery of the Leg: A Systematic Review and Meta-Analysis of Randomized Controlled Trials. J Am Heart Assoc. 2018 Dec 18;7(24):e011245. doi: 10.1161/JAHA.118.011245. PMID 30561254
- [Background] Clever YP, Peters D, Calisse J, Bettink S, Berg MC, Sperling C, Stoever M, Cremers B, Kelsch B, Bohm M, Speck U, Scheller B. Novel Sirolimus-Coated Balloon Catheter: In Vivo Evaluation in a Porcine Coronary Model. Circ Cardiovasc Interv. 2016 Apr;9(4):e003543. doi: 10.1161/CIRCINTERVENTIONS.115.003543. PMID 27069105
- [Background] Verheye S, Vrolix M, Kumsars I, Erglis A, Sondore D, Agostoni P, Cornelis K, Janssens L, Maeng M, Slagboom T, Amoroso G, Jensen LO, Granada JF, Stella P. The SABRE Trial (Sirolimus Angioplasty Balloon for Coronary In-Stent Restenosis): Angiographic Results and 1-Year Clinical Outcomes. JACC Cardiovasc Interv. 2017 Oct 23;10(20):2029-2037. doi: 10.1016/j.jcin.2017.06.021. Epub 2017 Sep 27. PMID 28964764
- [Background] Lok CE, Huber TS, Lee T, Shenoy S, Yevzlin AS, Abreo K, Allon M, Asif A, Astor BC, Glickman MH, Graham J, Moist LM, Rajan DK, Roberts C, Vachharajani TJ, Valentini RP; National Kidney Foundation. KDOQI Clinical Practice Guideline for Vascular Access: 2019 Update. Am J Kidney Dis. 2020 Apr;75(4 Suppl 2):S1-S164. doi: 10.1053/j.ajkd.2019.12.001. Epub 2020 Mar 12. PMID 32778223
- See also: Trends in Chronic Kidney Failure Stage 5 in Singapore 2013/2013 — https://www.nrdo.gov.sg/docs/librariesprovider3/Publications---Kidney-Failure/trends-in-chronic-kidney-failure-stage-5-in-singapore.pdf?sfvrsn=0
- See also: Updated CIRSE Position Statement on the use of Paclitaxel-Coated Balloons and Stents in Peripheral Arterial Disease. — https://www.radiologen.nl/sites/default/files/nieuws/cirse_position_statement.pdf